CLINICAL TRIAL: NCT06643793
Title: Evaluation of Irinotecan Liposome (II) Combined With 5-fluorouracil, Leucovorin, and Bevacizumab for Second-line/Third-line Treatment of Metastatic Colorectal Cancer (mCRC): a Prospective and Exploratory Clinical Study
Brief Title: Evaluation of Irinotecan Liposome (II) Combined With 5-FU, LV, and Bevacizumab for mCRC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Affiliated Hospital of Nantong University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRC-IIT-004
Record Dates: First submitted 2024-09-27; First posted 2024-10-16 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2024-09

CONDITIONS: Colorectal Neoplasms Malignant
MeSH Terms: conditions — Colonic Neoplasms | interventions — irinotecan sucrosofate; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Irinotecan liposome (Ⅱ) combined with 5-fluorouracil, leucovorin, and bevacizumab (Experimental): Irinotecan liposome (Ⅱ) + 5-FU/LV + bevacizumab
  Interventions: Drug: Irinotecan liposome (ll) + 5-FU/LV + bevacizumab

INTERVENTIONS:
Drug: Irinotecan liposome (ll) + 5-FU/LV + bevacizumab — 1. Bevacizumab: 5 mg/kg, d1, q2w;
  2. Irinotecan Hydrochloride Liposomal Injection (II): 60 mg/m2, d1, q2w;
  3. leucovorin: 400 mg/m2, d1, q2w;
  4. 5-fluorouracil: 2800 mg/m2, d1, q2w.

SUMMARY:
To observe and evaluate the efficacy and safety of irinotecan liposome (II) combined with 5-fluorouracil(5-FU), calcium leucovorin(LV), and bevacizumab in the treatment of metastatic colorectal cancer.

DETAILED DESCRIPTION:
Subjects enter the screening period after being fully informed and signing an informed consent form. The screening period for the study is 28 days. After completing the screening inspection and evaluation, the selected subjects receive irinotecan liposome (II) combined with 5-FU/LV and bevacizumab treatment, a total of 4 anti-tumor treatment cycles were observed. After the 4 cycles of treatment, the next step of treatment was jointly decided after the evaluation of the researcher and the consideration of the patient's personal treatment wishes.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old and ≤ 75 years old, gender is not limited;
2. Diagnosis of colorectal cancer by histopathology and/or cytology, clinical Records showing inoperable advanced metastatic colon or rectal cancer (ie, stage IV according to the UICC AJCC TNM staging system [8th edition 2017]) ;
3. At least 1 measurable target lesion according to RECIST v1.1 criteria (ie, non-nodal lesions with a CT scan length ≥10 mm and nodal lesions with a CT scan short diameter ≥15 mm) ;
4. Prior first- or second-line oxaliplatin-based therapy with treatment failure or intolerance*; Note: *Treatment failure or intolerance is defined as (1) disease progression during treatment or disease progression within 6 months of final treatment, both with clear evidence of imaging or clinical progression, and (2) patients who withdrew from treatment because of intolerance of an adverse event of the treatment, as per NCI-CTCAE v5.0 criteria, intolerance is defined as: a. Hematological toxicity: grade III neutropenia accompanied by fever >38.5°C, grade III thrombocytopenia with bleeding symptoms, and other grade IV or higher hematologic toxic reactions; b. Non-hematological toxicity: grade III or higher non-hematological toxic reactions; and c. Achievement of the above toxic reactions, which in the judgment of the investigator make continuation of the original regimen of Treatment.
5. ECOG physical status score 0-1;
6. Expected survival time ≥ 3 months;
7. No major organ dysfunction, that is, the subject's organ function level and related laboratory indicators must meet the following requirements within 14 days before the first medication: (1) Blood routine (no blood transfusion, platelet transfusion, growth factors and other supportive treatments): white blood cells (WBC) ≥ 3.0 × 109/L; Absolute neutrophil count (ANC) ≥ 1.5 × 109/L; Platelet count (PLT) ≥ 100 × 109/L; Hemoglobin (Hb) ≥ 90 g/L; (2) Blood biochemistry: serum albumin (ALB) ≥ 30 g/L; Alanine aminotransferase (ALT)/aspartate aminotransferase (AST) ≤ 2.5 times the upper normal value (ULN), and if there is liver metastasis, ALT/AST ≤ 5 × ULN; Total bilirubin (TBIL) ≤ 1.5 × ULN; Serum creatinine (Cr) ≤ 1.5 × ULN, or endogenous creatinine clearance ≥ 60 mL/min according to the Cockcroft-Gault formula; (3) Urine routine: urine routine indicates urine protein < + +; If the urinary protein at baseline is ≥ + +, it is necessary to confirm that the 24-hour urinary protein quantification is ≤ 1.0 g; (4) Coagulation function (within 14 days before the first dose): prothrombin time (PT) or activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN, international normalized ratio (INR) ≤ 1.5 × ULN (no anticoagulant therapy); If the subject is treated with a stable dose of anticoagulant or vitamin K antagonist (such as warfarin, heparin or their analogues), on the premise that the international normalized ratio (INR) of prothrombin time is ≤ 1.5, it is allowed to use low-dose warfarin (1 mg orally once a day) or low-dose aspirin (not exceeding 100 mg a day) for preventive purposes; (5) Cardiac function: normal 12-lead electrocardiogram or abnormal 12-lead electrocardiogram without clinical significance judged by the investigator (i.e., QTcF < 450 ms in men, QTcF < 470 ms in women); Left ventricular ejection fraction (LVEF) ≥ lower limit of normal value (i.e., LVEF ≥ 50%).
8. Other previous antineoplastic therapy should be terminated for 4 weeks or more, and the general physical condition or associated adverse effects have recovered (toxicity ≤1 grade) or reached a stable state;
9. Serum pregnancy test must be negative and non-lactation period in women of childbearing age within 7 days before receiving the test Women of child-bearing age or men whose partners are women of child-bearing age must agree to use medically approved contraception (e.g. , Intrauterine device, male surgical sterilization, birth control pills or condoms) for the duration of the trial;
10. Voluntarily participate and sign an informed consent form; Ability to comply with research visit plans and other program requirements.

Exclusion Criteria:

1. Have had a malignant tumor other than colorectal cancer within 5 years before the screening (cured skin basal cell or squamous cell carcinoma, cervical carcinoma in situ, and malignant tumors assessed by researchers as having a low risk of metastasis and death except);
2. Tumor tissue is known to have a mismatch repair defect (DMMR) status confirmed by immunohistochemistry, or a microsatellite high instability (MSI-H) status confirmed by second-generation sequencing (NGS) polymerase chain reaction (PCR) methods, they were evaluated by the investigators as being suitable for treatment with immune checkpoint inhibitors (PD-1/PD-L1 inhibitors)
3. The second generation sequencing (NGS)/polymerase chain reaction (PCR) method confirmed that it is a BRAF V600E mutation, which is unfavorable for patients with chemotherapy prognosis;
4. For those who are known to have central nervous system metastases, for patients with clinically suspected central nervous system metastases, enhanced computed tomography (CT) or enhanced nuclear magnetic resonance (MRI) must be performed within 28 days before the first medication to rule out central nervous system metastases;
5. Previous treatment with irinotecan/irinotecan liposome-based chemotherapy;
6. Use of CYP3A4, CYP2C8 and UGT1A1 strong inhibitors/strong inducers within 14 days before starting the study. 7. Participated in other drug clinical trials within 4 weeks before the first dose;
7. Participated in clinical trials of other drugs within 4 weeks before the first medication;
8. Clinical records showed severe gastrointestinal dysfunction (including bleeding and obstruction; NCI-CTCAE v5.0 > Grade 2 inflammation; NCI-CTCAE v5.0 > Grade 1 diarrhea)
9. Presence of severe comorbidities, active infections, or uncontrolled diabetes that interfere with the treatment of the trial drug: (1) uncontrolled severe medical disease that the investigators believe will affect the ability of the subject to receive treatment with the study regimen; For example, complicated with severe medical conditions, including severe heart disease, cerebrovascular disease, uncontrolled diabetes, uncontrolled hypertension, uncontrolled infection, active peptic ulcer, etc. (2) the occurrence of A/V thrombotic event within one year before screening, such as cerebrovascular accident (including transient ischemic attack) , thrombosis disease (except venous thrombosis caused by venous catheterization during pre-chemotherapy, which is judged to be cured by researchers) , pulmonary embolism, etc. (3) imaging showed that the tumor had invaded around the important blood vessels or the patients had a high possibility of invading the important blood vessels and causing fatal massive hemorrhage (4) the subjects had active, known or suspected autoimmune diseases including systemic lupus erythematosus, Hashimoto's thyroiditis, scleroderma, Polyarteritis nodosa or autoimmune hepatitis; Participants with type 1 diabetes, hypothyroidism requiring hormone replacement only, skin conditions that do not require systemic treatment (such as leukoplakia, psoriasis, or hair loss) , or conditions that are not expected to recur without an external trigger were allowed to participate; (5) active pulmonary tuberculosis infection. Patients with active tuberculosis infection within 1 year of treatment should be excluded, even if they have been treated, and patients with a history of active tuberculosis infection more than 1 year before should be excluded, (6) previous Interstitial lung disease, or has (non-infectious) pneumonia requiring oral or intravenous steroid hormone therapy; (7) long-term treatment with systemic sex hormones (at a dose equivalent to > 10 mg prednisone/day) or any other form of immunosuppressive therapy is required. Subjects who used inhaled or topical corticosteroid were selected, and those who had poorly controlled cardiac clinical symptoms or conditions, such as heart failure of NYHA Class 2 or above, unstable angina, and heart failure were selected Myocardial infarction within 6 months, clinically significant supraventricular or ventricular arrhythmias requiring treatment or intervention, positive Hepatitis C virus antibodies to HCV or HIV; Severe infection (NCI-CTCAE v5.0 > 2) occurred within 4 weeks before screening, such as severe pneumonia, bacteremia, infection complications, etc. The presence of symptoms and signs of infection within 2 weeks before study initiation required intravenous antibiotic therapy (except for prophylactic antibiotic use) ; (10) subjects with grade ≥2 peripheral neuropathy according to NCI-CTCAE v5.0.
10. Known to be allergic or intolerant to any test drug (irinotecan hydrochloride liposome injection (Ⅱ), 5-FU/LV, bevacizumab) or an excipient thereof;
11. There are known contraindications to any experimental drug (irinotecan hydrochloride liposome injection (Ⅱ), 5-FU/LV, bevacizumab);
12. Women who are pregnant, breastfeeding or have given birth but refuse to use contraception;
13. The researcher believes that it should be excluded from this study. For example, if the researcher judges that the subject has other factors that may lead to the forced termination of this study, such as the existence of other serious diseases (including mental illness) that require combined treatment, There are serious abnormalities in laboratory tests, accompanied by family or social factors, which will affect the safety of the subject or the collection of data and samples.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11-04 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 2 months after patient administration
  Investigator-assessed 2-month objective response rate (ORR) : proportion of subjects achieving a complete response (CR) or partial response (PR) in the analysis population according to RECIST v1.1 criteria 2 months after patient administration.

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | 2 months after patients administration
  Investigator-evaluated 2-month disease control rate (DCR): the proportion of subjects in the analysis population who achieved CR, PR or stable disease (SD) according to RECIST v1.1 criteria 2 months after patients administration
Treatment-related adverse events | 2 months after patient administration
  Evaluating the Safety of Investigational Drugs by NCI-CTC AE Version 5.0 Criteria

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Q Xue, Principal Investigator — Affiliated Hospital of Nantong University; Youlang Y Zhou, Principal Investigator — Affiliated Hospital of Nantong University; Feiran F Wang, Principal Investigator — Affiliated Hospital of Nantong University; Huajie H Miu, Principal Investigator — Affiliated Hospital of Nantong University
Locations (1):
- Affiliated Hospital Of Nantong University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No